CLINICAL TRIAL: NCT03695627
Title: Stress Free UCR: The Impact of 8 Weeks of Headspace on Stress in a Heterogeneous University Employee Cohort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Riverside (Other)
Collaborators: The University of California's Healthy Campus Network (Other); Headspace Meditation Limited (Industry); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Kate Sweeny, Professor of Psychology, University of California, Riverside
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-18-031
Record Dates: First submitted 2018-07-12; First posted 2018-10-04 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Stress, Psychological
Keywords: Stress, health, meditation, mindfulness, employees, job strain, burnout, work, help, mood, affect
MeSH Terms: conditions — Stress, Psychological; Occupational Stress; Burnout, Psychological; Helping Behavior | interventions — Meditation

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigator will be blind to condition throughout data accrual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation Group (Experimental): Participants in the meditation group will use a digitally-based mindfulness intervention Headspace app (Basics + Stress packs) will be used for 10 minutes a day over the course of 8 weeks
  Interventions: Behavioral: Meditation
- Control Group (No Intervention): Control group participants will continue their normal activities and not add any form of meditation during the study period.

INTERVENTIONS:
Behavioral: Meditation — 10 minute a day, 8 week digital meditation
  Arms: Meditation Group

SUMMARY:
The aim of this study is to test the effects of a digital meditation intervention in a sample of high stress UCR employees. We will randomize UCR employees to 8-weeks of either a digital mindfulness intervention (using the commercially available application Headspace) or a waitlist control condition.

Participants assigned to the intervention group will be asked to download and use the Headspace mobile application for 10 minutes per day for 8 weeks. They will be asked to fill out short (no longer than 30 minutes long) questionnaires at baseline, week 4, week 8 (post intervention), and a 4-month follow up period. Participants who are randomized to the digital meditation intervention will also take part in a 1-year follow up. All activities will take place online (via computer or smartphone), and on the participants' own time.

DETAILED DESCRIPTION:
High levels of psychosocial work-related stress have major implications for both the employee and the employer. Epidemiological studies consistently demonstrate associations between high work stress and worse self-reported mental and physical health, including depression, anxiety, cardiovascular disease, and type 2 diabetes.

Job strain, a combination of high demands and low control, is a common model used to define psychosocial stress at work. Job strain is associated with worse mental and physical health, including anxiety and depressive disorders and increased blood pressure.

Past studies show the value in mindfulness applications. For example, participants who completed 25 or more meditation sessions over 8 weeks also had significantly lower self-measured systolic blood pressure over the course of one day compared to the control condition participants at the follow-up time point. This trial suggests that almost daily brief mindfulness meditations delivered via smartphone can improve outcomes related to workplace stress and well-being, with potentially lasting effects.

In this study, investigators hope to determine if a stress-reduction mindfulness application is more effective than a waitlist control condition in employees who are experiencing mild to moderate levels of stress in various health and productivity-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Have access to a smartphone or computer every day
* Are fluent in English
* Are a UCR employee
* Have moderate to high levels of stress
* Consent: demonstrates understanding of the study and willingness to participate as evidenced by voluntary informed consent and has received a signed and dated copy of the informed consent
* Are at least 18 years of age

Exclusion Criteria:

* Experienced meditator or have participated in a formal meditation practice in the last 6 months (defined as 3-4 times or more per week)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Change in perceived stress score, as determined by the total score on the Perceived Stress Scale | Baseline to post-intervention, an anticipated average of 8 weeks
  The Perceived Stress Scale has a total score scale range of 0 to 40, with higher values indicating more perceived stress

SECONDARY OUTCOMES:
Change in subjective mindfulness, as determined by total score on Mindful Attention Awareness Scale | Baseline to post-intervention, an anticipated average of 8 weeks
  The Mindful Attention Awareness Scale is a 15-item measure with each item ranging from a score of 1 to 6. To score the scale, we compute the average score across items, with a higher score reflecting higher levels of mindfulness.
Anxiety, as determined by the Generalized Anxiety Disorder Scale | Baseline to post-intervention, an anticipated average of 8 weeks
  The Generalized Anxiety Disorder Scale is a 7-item measure with each item ranging from 0-3, with total scores ranging from 0-21 and higher scores indicating higher anxiety
Change in burnout, as determined by the Bergen Burnout Inventory | Baseline to post-intervention, an anticipated average of 8 weeks
  The Bergen Burnout Inventory is comprised of 9 items, ranging from 1 to 6. The total score range is from 9 to 54 with a higher score reflecting higher burnout.
Sleep quality as determined by the Pittsburgh Sleep Quality Index | Baseline to post-intervention, an anticipated average of 8 weeks
  The Pittsburgh Sleep Quality Index is a 9-item scale with a complex scoring scheme, in which a total score of "5" or greater is indicative of poor sleep quality
Worry as determined by the Penn State Worry Questionnaire | Baseline, 4 weeks, 8 weeks, 4 months, 1 year
  The Penn State Worry Questionnaire is a 16-item measure with total scores ranging from 16-60, and higher scores indicating more worry
Rumination as assessed by the McIntosh and Martin Rumination Questionnaire | Baseline, 4 weeks, 8 weeks, 4 months, 1 year
  The McIntosh and Martin Rumination Questionnaire is a 10-item measure with each item scored from 1-5, such that average scores range from 1 to 5 and higher scores indicate more rumination
Change in work engagement, as determined by the Utrecht Work Engagement Scale | Baseline to post-intervention, an anticipated average of 8 weeks
  The Utrecht Work Engagement scale is comprised of 9 items, with a total score ranging from 0 to 54, with higher scores indicating more work engagement.
Change in job strain, as determined by Siegrist Job Strain Scale | Baseline to post-intervention, an anticipated average of 8 weeks
  The job strain measure is a comprised of two sub scales, effort (5 items) and reward (11 items), each ranging from 1 to 4. The job strain score is calculated as the ratio of demand to reward, with a higher ratio reflecting more job strain.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Riverside, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ganster, D. C., & Rosen, C. C. (2013). Work stress and employee health. Journal of Management, 39(5), 1085-1122. https://doi.org/10.1177/0149206313475815
- [Background] Goh, J., Pfeffer, J., & Zenios, S. A. (2016). The Relationship Between Workplace Stressors and Mortality and Health Costs in the United States. Management Science, 62(2), 608-628. https://doi.org/10.1287/mnsc.2014.2115
- [Background] Karasek, R. A. (1979). Job Demands, Job Decision Latitude, and Mental Strain: Implications for Job Redesign. Administrative Science Quarterly, 24(2), 285. https://doi.org/10.2307/2392498
- [Background] Landsbergis PA, Dobson M, Koutsouras G, Schnall P. Job strain and ambulatory blood pressure: a meta-analysis and systematic review. Am J Public Health. 2013 Mar;103(3):e61-71. doi: 10.2105/AJPH.2012.301153. Epub 2013 Jan 17. PMID 23327240
- [Background] Landsbergis PA, Schnall PL, Warren K, Pickering TG, Schwartz JE. Association between ambulatory blood pressure and alternative formulations of job strain. Scand J Work Environ Health. 1994 Oct;20(5):349-63. doi: 10.5271/sjweh.1386. PMID 7863299
- [Background] Ly KH, Truschel A, Jarl L, Magnusson S, Windahl T, Johansson R, Carlbring P, Andersson G. Behavioural activation versus mindfulness-based guided self-help treatment administered through a smartphone application: a randomised controlled trial. BMJ Open. 2014 Jan 9;4(1):e003440. doi: 10.1136/bmjopen-2013-003440. PMID 24413342
- [Background] Mani M, Kavanagh DJ, Hides L, Stoyanov SR. Review and Evaluation of Mindfulness-Based iPhone Apps. JMIR Mhealth Uhealth. 2015 Aug 19;3(3):e82. doi: 10.2196/mhealth.4328. PMID 26290327
- [Background] Roeser, R. W., Schonert-Reichl, K. A., Jha, A., Cullen, M., Wallace, L., Wilensky, R., … Harrison, J. (2013). Mindfulness training and reductions in teacher stress and burnout: Results from two randomized, waitlist-control field trials. Journal of Educational Psychology, 105(3), 787-804. https://doi.org/10.1037/a0032093
- [Background] Siegrist J, Starke D, Chandola T, Godin I, Marmot M, Niedhammer I, Peter R. The measurement of effort-reward imbalance at work: European comparisons. Soc Sci Med. 2004 Apr;58(8):1483-99. doi: 10.1016/S0277-9536(03)00351-4. PMID 14759692
- [Background] The Sainsbury Centre for Mental Health. (2007). Mental Health at Work: Developing the business case (Vol. 8).
- [Background] Virgili, M. (2015). Mindfulness-based interventions reduce psychological distress in working adults: A meta-analysis of intervention studies. Mindfulness, 6(2), 326-337. https://doi.org/10.1007/s12671-013-0264-0
- [Background] Wolever RQ, Bobinet KJ, McCabe K, Mackenzie ER, Fekete E, Kusnick CA, Baime M. Effective and viable mind-body stress reduction in the workplace: a randomized controlled trial. J Occup Health Psychol. 2012 Apr;17(2):246-258. doi: 10.1037/a0027278. Epub 2012 Feb 20. PMID 22352291